CLINICAL TRIAL: NCT06666764
Title: Adjuvant Normobaric Hyperoxia in Acute Ischemic Stroke Patients Transferred for Thrombectomy
Brief Title: Normobaric Oxygen in AIS Transferred for EVT
Acronym: AN-O2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AN-O2
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; cerebral protection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO (Experimental): NBO will be conducted with inhalation of 100% oxygen. NBO will be used in conjunction with best medical practice.
  Interventions: Other: NBO
- Control (Other): Best medical treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: NBO — NBO will be conducted with inhalation of 100% oxygen.
  Arms: NBO
Other: Control — Best medical care
  Arms: Control

SUMMARY:
The primary objective of this study is to estimate the efficacy and safety of NBO on 3-month functional outcome after acute ischemic stroke

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability globally, with acute ischemic stroke (AIS) patients often benefiting from intravenous thrombolysis and endovascular therapies such as mechanical thrombectomy, which have been shown to improve reperfusion rates. However, despite reperfusion, the proportion of patients with large vessel occlusion achieving a favorable functional outcome, defined as a modified Rankin Scale score of 0-2 at 90 days, remains under 50%.

Normobaric hyperoxia (NBO) emerges as a compelling option for cerebral protection. Its neuroprotective mechanisms are thought to include hypoxic tissue rescue, blood-brain barrier preservation, brain edema reduction, neuroinflammation alleviation, mitochondrial function improvement, oxidative stress mitigation, and apoptosis inhibition. NBO's diffusion properties allow it to reach the penumbra before reperfusion, enhancing aerobic metabolism and potentially reducing infarct volume. Its advantages also include low cost, wide availability, and ease of use, making it accessible across various healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years old;
2. Signs and symptoms are consistent with a new acute stroke, with low possibility of stroke mimics (e.g., no sudden coma, prior seizure disorder, suspected hypoglycemia);
3. No prior stroke in the last 3 months;
4. Time from stroke onset (last seen well) to randomization is within 9 hours;
5. (1) Baseline NIHSS score at 6 or more and Intracranial ICA or MCA-M1 or MCA-M2 dominant occlusion, with or without tandem cervical carotid stenosis or tandem cervical occlusion, confirmed by preoperative CTA (or MRA, DSA) and consistent with signs and symptoms; or (2) Baseline NIHSS score at 6 or more with a hyperdense MCA sign on non-contrast CT; or (3) Baseline NIHSS score at 12 or more;
6. NIHSS score 0 or 1 in the section of level of consciousness;
7. No significant pre-stroke disability (pre-stroke mRS 0--1);
8. ASPECTS at least 6 on non-contrast CT;
9. Patient is planned for transfer to a EVT-capable hospital for EVT;
10. Signed informed consent from the patient or the legally authorized representative (LAR).

Exclusion Criteria:

1. Known history of severe chronic obstructive pulmonary disease (FEV1 less than 1.0), New York Heart Association (NYHA) Heart Failure Class III or IV, acute pulmonary infection or aspiration pneumonia, prior to enrollment;
2. Respiratory rate <= 10 or >= 30 breaths per minute;
3. Oxygen-dependence at baseline to maintain SaO2 > 95% or intubation at baseline;
4. Seizure at stroke onset;
5. Exhibiting symptoms of vomiting, or severe headache, or unconscious;
6. Rapidly improving neurological deficits or transient ischemic attack prior to consent;
7. Signs and symptoms suggestive of subarachnoid hemorrhage, even if CT scan is normal;
8. Evidence of intracranial tumor (except small meningioma) or arteriovenous malformation;
9. Woman of childbearing potential known to be pregnant or with a positive pregnancy test;
10. Life expectancy < 90 days due to comorbidity;
11. Unlikely to complete the 90-day follow-up;
12. Participating in another clinical treatment trial, or completed participation within prior 30 days;
13. Receiving other cerebral protective agent (e.g., edaravone dexborneol, n-butylphthalide);
14. Evidence of acute intracranial hemorrhage on CT/MRI;
15. Significant mass effect with midline shift, defined as any deviation of midline structures such as the septum pellucidum, is observed on CT/MRI scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Level of disability measured by modified Rankin scale (mRS) score | 90 days, 1 year after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome; the primary outcome here is 3-month ordinal mRS score with mRS 5 and 6 merged into one category; modified intention-to-treat analysis

SECONDARY OUTCOMES:
Functional independence defined as the proportion of patients with a modified Rankin scale (mRS) score of 0-2 at follow up | 90 days, 1 year after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome. The mRS score is dichotomized to define the functional independence as mRS score of 0-2.
Excellent functional outcome, defined as the proportion of patients with a modified Rankin scale (mRS) score of 0-1 at follow up | 90 days, 1 year after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome. The mRS score is dichotomized to define the excellent functional outcome as mRS score of 0-1.
National Institutes of Health Stroke Scale (NIHSS) | 24 hours after randomization
  The National Institutes of Health Stroke Scale (NIHSS) ranges from 0 to 42 points, with higher scores indicating worse neurological deficits.
Early neurological improvement | 24 hours after randomization
  Neurological improvement is defined as a decrease of at least 4-point reduction in NIHSS score at 24 hours of randomization to baseline assessment
Alberta Stroke Program Early CT (ASPECT) score upon the Endovascular Thrombectomy (EVT) sites' admission | Day 0, Endovascular Thrombectomy (EVT) site admission
  Alberta Stroke Program Early CT (ASPECT) score ranges from 0 to 10, with 10 being normal and 0 indicating complete MCA infarction
Change of Infarct volume at 24 hours from baseline | 24 (+/- 12) hours after randomization
  Both the infarct volume at 24 hours and the change of it from baseline will be analyzed
EuroQol five dimensions questionnaire（EQ-5D） | 90 days, 1 year after randomization
  The score ranges from 0 to 100, with higher scores indicating optimal health
Excellent functional outcome at day 5 (or discharge if earlier) defined as modified ranking scale (mRS) score of 0-1 at day 5 (or discharge if earlier) | Day 5 (or discharge if earlier) after randomization
  The original modified ranking scale (mRS) score ranges from 0 to 6, with higher scores indicating a worse outcome. We use the dichotomozed mRS score to define the excellent functional outcome as mRS score of 0-1 at day 5 (or discharge if earlier).
Functional independence at day 5 (or discharge if earlier) defined as modified ranking scale (mRS) score of 0-2 at day 5 (or discharge if earlier) | Day 5 (or discharge if earlier) after randomization
  The original modified ranking scale (mRS) score ranges from 0 to 6, with higher scores indicating a worse outcome. We use the dichotomozed mRS score to define the functional independence as mRS score of 0-2 at day 5 (or discharge if earlier).
Spontaneous or IV thrombolysis induced recanalization from baseline to Endovascular Thrombectomy (EVT) site arrival | Day 0, Endovascular Thrombectomy (EVT) site admission
  Among patients who have related imaging from both the non-EVT and EVT sites
Barthel Index | 90 days, 1 year after randomization
  The Barthel Index is an ordinal disability score of 10 categories (range from 0 to 100, higher values indicate better prognosis)

OTHER OUTCOMES:
Serious adverse events/Adverse events | Through study completion
  total number of serious adverse events/adverse events reported during follow-up, according to standard definitions
Symptomatic intracranial hemorrhage | Up to 36 hours after randomization
  Number of cases of symptomatic intracerebral hemorrhage according to standard definition
Any intracranial hemorrhage | Up to 36 hours after randomization
  Number of cases of any intracranial hemorrhage according to standard definitions
Early neurological deterioration | 24 hours after randomization
  Early neurological deterioration at 24 hours, defined as at least 4-point increase in NIHSS score from baseline;
Vital signs | Day 0, at the end of oxygen therapy
  Vital signs at the end of oxygen therapy, including heart rate, respiratory rate, systolic blood pressure, diastolic blood pressure, and oxygen saturation

CONTACTS AND LOCATIONS:
Locations (112):
- China (112):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University First Affiliated Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Minhou County Hospital, Fuzhou, Fujian
  - Fuqing Hospital, Fuzhou, Fujian
  - Fuqing Second Hospital, Fuzhou, Fujian
  - Fuzhou Changle District People's Hospital, Fuzhou, Fujian
  - Fuzhou Traditional Chinese Medicine Hospital, Fuzhou, Fujian
  - Lianjiang County General Hospital, Fuzhou, Fujian
  - Luoyuan County Hospital, Fuzhou, Fujian
  - Minqing County General Hospital, Fuzhou, Fujian
  - Yongtai County Hospital, Fuzhou, Fujian
  - Gutian County Hospital, Ningde, Fujian
  - Putian Hanjiang District Hospital, Putian, Fujian
  - Dongshan County Hospital, Zhangzhou, Fujian
  - Nanjing County Hospital, Zhangzhou, Fujian
  - Pinghe County Hospital, Zhangzhou, Fujian
  - Xiage Health Center, Zhangzhou, Fujian
  - Yunxiao County Hospital, Zhangzhou, Fujian
  - Yunxiao County Traditional Chinese Medicine Hospital, Zhangzhou, Fujian
  - Zhangpu County Hospital, Zhangzhou, Fujian
  - Zhangpu County Traditional Chinese Medicine Hospital, Zhangzhou, Fujian
  - Zhangzhou Changtai District Hospital, Zhangzhou, Fujian
  - Zhangzhou Fifth Hospital, Zhangzhou, Fujian
  - Zhangzhou Gulei Port Economic Development Zone First Hospital, Zhangzhou, Fujian
  - Zhangzhou Hospital Headquarters (High-Tech Campus), Zhangzhou, Fujian
  - Zhangzhou Hospital, Zhangzhou, Fujian
  - Zhangzhou Second Hospital, Zhangzhou, Fujian
  - Zhao'an County Hospital, Zhangzhou, Fujian
  - Guangzhou Development District Hospital, Guangzhou, Guangdong
  - Guangzhou He Xian Memorial Hospital, Guangzhou, Guangdong
  - Jinan University First Affiliated Hospital, Guangzhou, Guangdong
  - Yifeng County People's Hospital, Guangzhou, Guangdong
  - Fuchuan Yao Autonomous County Ethnic Medicine Hospital, Hezhou, Guangxi
  - Hezhou Traditional Chinese Medicine Hospital, Hezhou, Guangxi
  - Zhaoping County People's Hospital, Hezhou, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Dongguang County People's Hospital, Cangzhou, Hebei
  - Xianxian Traditional Chinese Medicine Hospital, Cangzhou, Hebei
  - Daming County Traditional Chinese Medicine Hospital, Handan, Hebei
  - Handan Central Hospital (East Campus), Handan, Hebei
  - Handan Fourth Hospital, Handan, Hebei
  - Linzhang County People's Hospital, Handan, Hebei
  - Quzhou County Hospital, Handan, Hebei
  - Linkou County People's Hospital, Mudanjiang, Heilongjiang
  - Mudanjiang Second People's Hospital, Mudanjiang, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - Song County People's Hospital, Luoyang, Henan
  - Xin'an County People's Hospital, Luoyang, Henan
  - Yichuan County People's Hospital, Luoyang, Henan
  - Yima People's Hospital, Yima, Henan
  - Yimei General Hospital, Yima, Henan
  - Danchuan County Traditional Chinese Medicine Hospital, Zhoukou, Henan
  - Luyi Zhenyuan Hospital, Zhoukou, Henan
  - Shenqiu County People's Hospital, Zhoukou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Danchuan Central Hospital, Zhoukou, Hennan
  - Hubei Minzu University Affiliated Minzu Hospital, Enshi, Hubei
  - Huangmei County People's Hospital, Huanggang, Hubei
  - Lichuan Traditional Chinese Medicine Hospital, Lichuan, Hubei
  - Dexing People's Hospital, Dexing, Jiangxi
  - Guangchang County People's Hospital, Fuzhou, Jiangxi
  - Jinxi County People's Hospital, Fuzhou, Jiangxi
  - Zixi County People's Hospital, Fuzhou, Jiangxi
  - Dean County People's Hospital, Jiujiang, Jiangxi
  - Dean County Traditional Chinese Medicine Hospital, Jiujiang, Jiangxi
  - Hukou County People's Hospital, Jiujiang, Jiangxi
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - Pengze County People's Hospital, Jiujiang, Jiangxi
  - Xiajiang County People's Hospital, Ji’an, Jiangxi
  - Xingan County People's Hospital, Ji’an, Jiangxi
  - Yongfeng County Traditional Chinese Medicine Hospital, Ji’an, Jiangxi
  - Lushan People's Hospital, Lushancun, Jiangxi
  - Anyi County People's Hospital, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Xinjian District People's Hospital, Nanchang, Jiangxi
  - Poyang County People's Hospital, Shangrao, Jiangxi
  - Wannian County People's Hospital, Shangrao, Jiangxi
  - Fengxin County People's Hospital, Yichun, Jiangxi
  - Shanggao County People's Hospital, Yichun, Jiangxi
  - Yujiang District People's Hospital, Yingtan, Jiangxi
  - Zhangshu People's Hospital, Zhangshu, Jiangxi
  - Baoji High-Tech Hospital, Baoji, Shaanxi
  - Caijiapo Hospital, Baoji, Shaanxi
  - Longxian People's Hospital, Baoji, Shaanxi
  - Meixian Traditional Chinese Medicine Hospital, Baoji, Shaanxi
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Feicheng Hospital of Shandong Yiyang Health Group, Tai’an, Shandong
  - Jincheng First People's Hospital, Jinzhong, Shanxi
  - Xiyang County People's Hospital, Jinzhong, Shanxi
  - Wenshui County People's Hospital, Lüliang, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Binchuan County People's Hospital, Dali, Yunnan
  - Binchuan County Traditional Chinese Medicine Hospital, Dali, Yunnan
  - Dali Prefecture People's Hospital, Dali, Yunnan
  - Heqing County People's Hospital, Dali, Yunnan
  - Jianchuan County People's Hospital, Dali, Yunnan
  - Midu County People's Hospital, Dali, Yunnan
  - Nanjian Yi Autonomous County People's Hospital, Dali, Yunnan
  - Yangbi County People's Hospital, Dali, Yunnan
  - Yongping County People's Hospital, Dali, Yunnan
  - Chenggong District People's Hospital, Kunming, Yunnan
  - Jinning District People's Hospital, Kunming, Yunnan
  - Kunming Medical University Yan'an Hospital, Kunming, Yunnan
  - Songming County People's Hospital, Kunming, Yunnan
  - Yiliang First People's Hospital, Kunming, Yunnan
  - Yunnan Provincial First People's Hospital, Kunming, Yunnan
  - The First People's Hospital of Qujing, Qujing, Yunnan
  - Fuyuan County People's Hospital, Qujing, Yunnan
  - Shizong County People's Hospital, Qujing, Yunnan
  - Xuanwei First People's Hospital, Xuanwei, Yunnan
  - Yuxi Zhongshan Hospital, Yuxi, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided